CLINICAL TRIAL: NCT06844669
Title: HER2HEART-US: Primary Prevention of Cardiotoxicity in Breast Cancer Patients Receiving HER2-directed Therapy: a Pilot 2x2 Factorial Randomized Controlled Trial
Brief Title: HER2HEART-US: Prevention of Cardiotoxicity in Breast Cancer Patients Receiving HER2-directed Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 202502113
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Breast Cancer; HER2+ Breast Cancer
Keywords: Breast cancer; Cardiotoxicity; Heart failure; Cardio-oncology
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Heart Failure | interventions — Carvedilol; empagliflozin

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial, open-label, randomized pilot study. Patients will be randomized on a 1:1 basis to either carvedilol or no carvedilol, and again on a 1:1 basis to either empagliflozin or no empagliflozin, meaning that there are four arms:
  * Arm 1: carvedilol
  * Arm 2: empagliflozin
  * Arm 3: carvedilol + empagliflozin
  * Arm 4: usual care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Carvedilol BID (Experimental): Carvedilol by mouth twice per day (BID) for 12 weeks.
  Interventions: Drug: Carvedilol
- Arm 2: Empagliflozin QD (Experimental): Empagliflozin by mouth daily (QD) for 12 weeks.
  Interventions: Drug: Empagliflozin
- Arm 3: Carvedilol BID + Empagliflozin QD (Experimental): Carvedilol by mouth twice per day (BID) for 12 weeks and empagliflozin by mouth daily (QD) for 12 weeks.
  Interventions: Drug: Carvedilol; Drug: Empagliflozin
- Arm 4: Usual Care (No Intervention): No medications.

INTERVENTIONS:
Drug: Carvedilol — 6.25 mg with food
  Other Names: Coreg
  Arms: Arm 1: Carvedilol BID; Arm 3: Carvedilol BID + Empagliflozin QD
Drug: Empagliflozin — 10 mg in the morning with or without food
  Other Names: Jardiance
  Arms: Arm 2: Empagliflozin QD; Arm 3: Carvedilol BID + Empagliflozin QD

SUMMARY:
Ten to 15% of patients with breast cancer are HER2 positive, with treatment focused on targeting the HER2 receptor. Although these treatments are generally well tolerated, they are associated with an increased risk of cardiomyopathy. There are currently no treatments proven to prevent the cardiotoxicities associated with HER2-targeted therapy, but there is convincing preclinical data demonstrating that prophylactic treatment with a beta blocker (BB) and/or an SGLT2 inhibitor (SGLT2i) may each independently prevent cardiotoxicity and HER-targeted treatment interruptions.

The proposed pilot study will assess the feasibility and preliminary efficacy and safety of therapy with both a beta blocker (carvedilol) and an SGLT2 inhibitor (empagliflozin), alone and in combination, in a population initiating HER2-directed therapy for HER2+ breast cancer.

The hypotheses being tested in this study are:

1. It is feasible to recruit 20-40 patients over 6 months
2. There are no differences in tolerability and safety between participants taking carvedilol and/or empagliflozin and those receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2+ breast cancer by ASCO/CAP guidelines of any clinical or pathologic stage.
* Planning to commence standard of care HER2-directed therapy or started HER2-directed therapy within 6 months prior to randomization
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* For patients newly commencing HER2-directed therapy, left ventricular ejection fraction (LVEF) ≥ 50% up to 30 days prior to enrollment detected by echocardiogram. For patients already receiving HER2-directed therapy, LVEF ≥ 50% after the last cycle of therapy prior to enrollment. (Patient will be enrolled at the time of their next cycle after the echocardiogram.)
* Systolic blood pressure ≥ 100 mmHg and resting heart rate ≥ 60 bpm.
* eGFR > 30 mL/min/1.73m^2.
* Women of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patients with an acceptable support system (as determined by the treating medical team).
* Ability to understand and willingness to sign an Institutional Review Board (IRB) approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior exposure to mantle cell lymphoma field radiation.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen as determined by the treating physician. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving treatment with SGLT2i or BB that cannot be stopped during the duration of study participation. Currently receiving non-dihydropyridine calcium channel blocker that cannot be transitioned to or used in combination with carvedilol.
* Patients with untreated brain metastases requiring central nervous system directed therapy and interruption of systemic HER2 directed therapy (as determined by the treating medical team.
* A known history of allergic reactions attributed to compounds of similar chemical or biologic composition to carvedilol, empagliflozin, or other agents used in the study.
* Contraindication to carvedilol or empagliflozin at the discretion of the investigator such as:

  * Bronchial asthma or related bronchospastic conditions where BB would be contraindicated
  * Second- or third-degree atrioventricular (AV) block
  * Sick sinus syndrome
  * Severe bradycardia (unless permanent pacemaker in place)
  * In cardiogenic shock or decompensated heart failure requiring the use of IV inotropic therapy
  * Severe hepatic impairment in setting of cirrhosis that prevents use of carvedilol
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection or uncontrolled cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of HER2HEART as measured by the number of patients enrolled over a 10-month period | 10 months
  Feasibility is defined as enrollment of 20-40 patients (5-10 per am) over a 10-month recruitment period.

SECONDARY OUTCOMES:
Tolerability as measured by treatment adherence via self-report | From start of treatment through last day of study treatment (estimated to be 3 months)
Tolerability as measured by incidence of serious adverse events | From start of treatment through last day of study treatment (estimated to be 3 months)
Tolerability as measured by incidence of adverse events of special interest | From start of treatment through last day of study treatment (estimated to be 3 months)
  * Symptomatic hypotension (systolic blood pressure <90 mmHg)
  * Symptomatic bradycardia (heart rate <50 bpm)
  * Acute renal dysfunction (eGFR decrease >30% from baseline)
  * Syncope
  * Symptomatic hypoglycemia (blood glucose <70 mg/dL)
  * Perineal infection
  * Urinary tract infection
  * Diabetic ketoacidosis (commonly accepted criteria are blood glucose > 250 mg/dL, arterial pH < 7.3, serum bicarbonate < 15 mEq/L, and the presence of ketonemia or ketonuria).
  * Euglycemic diabetic ketoacidosis (diabetic ketoacidosis in the absence of hyperglycemia)
Tolerability as measured by number of participants who withdraw from the study due to adverse events | From start of treatment through last day of study treatment (estimated to be 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mitchell, M.D., MSCI, FAC, FICOS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared after deidentification. These requests are reviewed and will be approved by study investigators on the basis of scientific merit.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication.
Access Criteria: These requests are reviewed and will be approved by study investigators on the basis of scientific merit.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu